CLINICAL TRIAL: NCT06089473
Title: Virtual Home-based Physical Pre-habilitation in Kidney Transplant Candidates: a Pilot RCT
Brief Title: Virtual Home-based Physical Pre-habilitation in Kidney Transplant Candidates
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: The Kidney Foundation of Canada (Other)
Responsible Party: Principal Investigator, Tania Janaudis-Ferreira, Scientist, Translational Research in Respiratory Diseases Program, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023-10799
Record Dates: First submitted 2023-10-05; First posted 2023-10-18 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Kidney Disease, End-Stage; Frailty; Transplant;Failure,Kidney
MeSH Terms: conditions — Kidney Failure, Chronic; Frailty | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: RCT with 2 arms
Who Masked: Outcomes Assessor
Masking Description: outcomes will be assessed without knowledge of group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Pre-habilitation plus usual outpatient care (Other): An intervention including exercise and education.
  Interventions: Other: Intervention Group: Exercise and education.
- No Intervention: Usual outpatient care (Other): The control group will receive usual outpatient care provided to kidney transplant candidates. All participants in the control group will receive educational resources received by intervention group participants at trial completion.
  Interventions: Other: Usual Care Only

INTERVENTIONS:
Other: Intervention Group: Exercise and education. — * Exercise Intervention: 12-weeks of supervised, individualized virtual exercise sessions, delivered by an accredited kinesiologist. Independent unsupervised sessions start at week 5. After 12 weeks, a 5-month maintenance phase is followed, continuing to exercise three times weekly for 30 minutes per session.
  * Education: Prior to each zoom session with the kinesiologist (starting on week 2), participants will watch short educational videos. Additionally, participants will be provided a document (PDF) of evidence-based strategies to help cope with stress.
  Arms: Experimental: Pre-habilitation plus usual outpatient care
Other: Usual Care Only — Usual Care for kidney transplant candidates, which may include medical visits, nutrition, and psychological support.
  Arms: No Intervention: Usual outpatient care

SUMMARY:
The goal of this RCT is to address the feasibility of conducting a 12-week virtual pre-habilitation intervention, which includes exercise and education, in kidney transplant candidates. The intervention also includes a 5-month maintenance phase with independent home exercises (maximum of 8 months of intervention/ended early if the participant undergoes a kidney transplant). The main questions it aims to answer are:

* estimate the proportion of screened patients who meet eligibility criteria
* estimate the proportion of eligible patients who consent to randomization
* estimate the proportion of patients who adhere to the interventions
* estimate follow-up completion rates
* inform the calculation of sample size requirements for a full-scale RCT
* assess the acceptability of the intervention by the participants.

Participants in the control group will receive usual outpatient care.

DETAILED DESCRIPTION:
While waiting for kidney transplant, candidates face many challenges related to their physical health. These physical impairments are strongly associated with pre- and post-transplant mortality and morbidity. Pre-habilitation is the process of enhancing patient functional capacity prior to surgery with the objective of improving tolerance for the stressor. In the context of this protocol, pre-habilitation is referring to an exercise-based program with education prior to transplant. Pre-habilitation has been shown to contribute to a reduction of postoperative recovery time and quicker return to functional ability after thoracic and abdominal surgery. There is, however, limited evidence for the effects of pre-habilitation in kidney transplant candidates.

The investigators are following up previous work conducted with a very small (n=8) pilot pre-post study on pre-habilitation (MUHC REB number = 2020-5951) specifically with kidney transplant candidates. The results were encouraging.

The current multicenter pilot randomized controlled trial (RCT) will address the following research question: is it feasible to conduct a full-scale multicenter RCT to assess the comparative effectiveness of a virtual home-based pre-habilitation versus usual care for kidney transplant candidates? The investigators' specific objectives are to: (1) estimate the proportion of screened patients who meet eligibility criteria, (2) estimate the proportion of eligible patients who consent to randomization, (3) estimate the proportion of patients who adhere to the interventions, (4) estimate follow-up completion rates, (5) inform the calculation of sample size requirements for a full-scale RCT and, (6) assess the acceptability of the intervention by the participants. The assessor-blind pilot RCT will be conducted in three hospitals in Canada: MUHC, CHUM and University of Alberta Hospital. Eligible subjects will be randomized 1:1 to receive either i) virtual home-based multimodal pre-habilitation plus usual outpatient care, or ii) usual outpatient care. Participants will be drawn from the transplant clinics at the 3 sites, and the investigators aim to recruit 30 participants (22 of which will be recruited from MUHC over 9 months).

While some of the assessment appointments will be in person, the intervention is virtual so as not to burden the participants with extra hospital visits. The exercise portion of the study will include a 12-week virtual home-based supervised exercise program and a 5-month maintenance phase with independent home exercises (maximum of 8 months of intervention/ended early if the participant undergoes transplantation). Participants in the intervention group will also watch short educational videos about their kidney, assessment and waitlist, surgery and recovery, medication, and their new life after transplantation. Additionally, participants will be provided a document (PDF) of evidence-based strategies to help cope with stress.

Patients in the control group will receive usual outpatient care. All participants in the control group will receive educational resources received by intervention group participants at trial completion.

All participants will undergo a nutrition screening and will complete questionnaires regarding anxiety and depression. The corresponding transplant team will be notified should participants score 'abnormal' on these assessment tools. Additionally, all study participants will be asked questions regarding the following: whether they have had previous nutritional counselling or received any nutritional interventions, whether they have nutritional concerns/needs, whether they face any challenges in maintaining a balanced diet, whether they have had previous psychological counseling as part of the transplant assessment. This information will be collected as part of a needs assessment to inform inclusion of a nutritional and psychological interventions in subsequent trials.

ELIGIBILITY:
Inclusion Criteria:

* consecutive individuals with end stage kidney disease (ESKD) (aged ≥18 years), classified as pre-frail (1-2 points), frail (3-4 points) or very frail (5 points) on the Fried's frailty phenotype and who are accepted or in the process of being accepted to enter in the deceased or living donor KT waiting list of the McGill University Health Centre (MUHC), Centre Hospitalier de l'Université de Montreal (CHUM) or University of Alberta Hospital (UAH) for first-time transplantation or re-transplantation
* English or French speakers
* is technologically capable of connecting (either independently or through household members/next-of-kin) with an online videoconferencing platform through an e-mail invitation (Patients who do not have access to internet will borrow a tablet with internet for the period of the study)

Exclusion Criteria:

* Individuals who:
* are classified as robust (0 points) on their Fried's frailty phenotype score
* are participating in a structured exercise program (hospital-based or home-based or another trial)
* are waiting for kidney-pancreas or kidney-liver transplant as those have much longer waiting time
* are hospitalized for any reason during the assessment for eligibility
* have a cPRA (calculated panel reactive antibodies) >95% and are on the highly sensitized exchange program and expected to have a prolonged waiting times on the waiting list
* are expected to have a transplant before the end of the 12 week-intervention (e.g. individuals who will receive an organ from a living donor or are type A blood
* have pre-existing or newly identified significant cognitive impairment
* have pre-existing or newly identified cardiac, musculoskeletal, neuropathy or neurological condition that might affect their exercise performance or otherwise render rehabilitation participation unsafe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-02 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of screened patients who meet eligibility criteria | at 12 months
  Data generated from this pilot RCT will inform the feasibility of a full-scale RCT by testing the study procedures; therefore, no inferential statistical analyses will be performed to compare groups. Socio-demographic, anthropometric and clinical data will be described using means and standard deviation or median and interquartile range for continuous variables and number and percentage for categorical variables. The variables will be presented at baseline, end of the 12 weeks (induction phase), at 6 months (during maintenance phase), at 8 months (end of maintenance phase) at 3-month post-transplant. Descriptive statistics (frequencies and percentages) will be used to report the feasibility and safety outcomes.
Proportion of eligible patients who consent to randomization | at 12 months
  Data generated from this pilot RCT will inform the feasibility of a full-scale RCT by testing the study procedures; therefore, no inferential statistical analyses will be performed to compare groups. Socio-demographic, anthropometric and clinical data will be described using means and standard deviation or median and interquartile range for continuous variables and number and percentage for categorical variables. The variables will be presented at baseline, end of the 12 weeks (induction phase), at 6 months (during maintenance phase), at 8 months (end of maintenance phase) at 3-month post-transplant. Descriptive statistics (frequencies and percentages) will be used to report the feasibility and safety outcomes.
Proportion of patients who adhere to the interventions | at 12 months
  Data generated from this pilot RCT will inform the feasibility of a full-scale RCT by testing the study procedures; therefore, no inferential statistical analyses will be performed to compare groups. Socio-demographic, anthropometric and clinical data will be described using means and standard deviation or median and interquartile range for continuous variables and number and percentage for categorical variables. The variables will be presented at baseline, end of the 12 weeks (induction phase), at 6 months (during maintenance phase), at 8 months (end of maintenance phase) at 3-month post-transplant. Descriptive statistics (frequencies and percentages) will be used to report the feasibility and safety outcomes.
Rate of follow-up completion as assessed by number of randomized patients completing assessments pre- and post-induction phase. | at 12 months
  Data generated from this pilot RCT will inform the feasibility of a full-scale RCT by testing the study procedures; therefore, no inferential statistical analyses will be performed to compare groups. Socio-demographic, anthropometric and clinical data will be described using means and standard deviation or median and interquartile range for continuous variables and number and percentage for categorical variables. The variables will be presented at baseline, end of the 12 weeks (induction phase), at 6 months (during maintenance phase), at 8 months (end of maintenance phase) at 3-month post-transplant. Descriptive statistics (frequencies and percentages) will be used to report the feasibility and safety outcomes. Completeness to follow-up will be compared between trial arms.

SECONDARY OUTCOMES:
Rate of change in frailty status as assessed by Fried's phenotype method | At baseline, post-induction phase (12 weeks), at 6 months, at 8 months, at 3-month post-transplant
  Frailty status as measured at the timepoints described below will use the Fried's phenotype method, identified by 3 or more of the following criteria.
  (please see each component outlined as its own outcome measure).
  1. Weight loss
  2. Weakness will be assessed using the handgrip strength test ith cut-off values provided by the Frailty index to determine weakness.
  3. Exhaustion:
  4. Slow gait:
  5. Low physical activity:
  Scoring for the Fried Phenotype: Each indicator can have 0 or 1 as a score, resulting in a total of maximum 5 points, where 0 is being robust, 1-2 pre-frail, 3-4 frail and 5 very frail.
Rate of change in bodyweight obtained from electronic medical chart (contributing to frailty status score for Fried's phenotype method). | At baseline, post-induction phase (12 weeks), at 6 months, at 8 months, at 3-month post-transplant
  Weight loss (of > 10 lbs over 6 months): obtained from the patient or chart.
Rate of change in handgrip strength as assessed by hand dynamometer (contributing to frailty status score for Fried's phenotype method). | At baseline, post-induction phase (12 weeks), at 6 months, at 8 months, at 3-month post-transplant
  Weakness will be assessed using the handgrip strength test (Jamar hydraulic hand Dynamometer). Patients will do six measurements (three times for each hand, with a rest break of 30 seconds between each). The highest measurement will be compared with cut-off values provided by the Frailty index to determine weakness.
Incidence of exhaustion as assessed by Center for Epidemiological Studies Depression (CES-D) (contributing to frailty status score for Fried's phenotype method). | At baseline, post-induction phase (12 weeks), at 6 months, at 8 months, at 3-month post-transplant
  Exhaustion will be measured by self-reported information based on two questions relating to feeling unusually tired and/or weak, taken from the Center for Epidemiological Studies Depression (CES-D) scale.
Rate of change in gait speed as assessed by the 4-metre gait speed test (contributing to frailty status score for Fried's phenotype method). | At baseline, post-induction phase (12 weeks), at 6 months, at 8 months, at 3-month post-transplant
  Slow gait: the 4-meter gait speed test will be used to analyze walking time. Participants will be timed as they walk 4 metres at their usual walking pace.
Rate of change in low physical activity status as assessed by the Rapid Assessment of Physical Activity (RAPA) questionnaire (contributing to frailty status score for Fried's phenotype method). | At baseline, post-induction phase (12 weeks), at 6 months, at 8 months, at 3-month post-transplant
  Low physical activity: energy expenditure weekly rate calculated using the Rapid Assessment of Physical Activity (RAPA) questionnaire; its 7 items assess habits of volume and intensity of weekly exercise. The score will determine whether participants are active or under-active. The scale ranges from 1 (sedentary) to 7 (active). A score of 5 (under-active regular) or less qualifies as low physical activity.
Rate of change in lower-extremity function will be assessed using the short physical performance battery (SPPB). | At baseline, post-induction phase (12 weeks), at 6 months, at 8 months, at 3-month post-transplant
  The short physical performance battery (SPPB) includes 3 brief physical fitness tests contributing to an overall score demarcating level of frailty. The tests include a 4-metre usual pace walk, a five-repetition sit-to-stand test, and balance tests.
Rate of change in functional exercise capacity as assessed by the 6-minute walk test | At baseline, post-induction phase (12 weeks), at 6 months, at 8 months, at 3-month post-transplant
  Functional exercise capacity will be measured using the 6-minute walking test (6MWT), which uses the distance walked within 6 minutes in metres. The 6MWT has been shown to be a reliable and viable alternative to the gold standard test (cardiopulmonary exercise test) in individuals with chronic kidney disease.
Rate of change in Health Related Quality of Life scores as assessed by the Kidney Disease Quality of Life Short Form Instrument (KDQOL-SF) | At baseline, post-induction phase (12 weeks), at 6 months, at 8 months, at 3-month post-transplant
  Kidney Disease Quality of Life Short Form Instrument (KDQOL-SF) is a self-report measure developed for individuals with kidney disease and those on dialysis. It includes both generic (36 items) and disease-specific (43 items) components for the assessment of HRQoL. Life Participation will be assessed using sub-scales of the KDQOL-SF questionnaire which include questions about personal relationships, work, and activities of daily living. The minimum and maximum scores vary by question, as does the scoring for those items. In some of the items, a higher numerical score (5/5) indicates a favourable health state, whereas the opposite is true for other items (1/5) indicates a more favourable health state. The scoring procedure for the KDQOL-SF transforms the numeric values into a 1-100 range, with higher transformed scores reflecting a better quality of life.
Changes in nutrition status as assessed by Patient-Generated Subjective Global Assessment (PG-SGA) | For those who receive a transplant within study period: baseline and 3-months post-transplant. For those who do not receive a transplant during study period: baseline and 8-months.
  Patient-Generated Subjective Global Assessment (PG-SGA) Scale Information: this is a patient-scored questionnaire in which participants will note changes in food intake, appetite changes, and activity levels. This scale ranges from 0 (no problems) to 36 (worst problem), with a higher score reflecting a greater risk for malnutrition. A score of 9 or above indicates a need for nutritional intervention.
Rate of change in body composition as measured by Bioelectrical Impedance | At baseline, post-induction phase (12 weeks), at 6 months, at 8 months, at 3-month post-transplant.
  Bioelectrical impedance will measure measure body composition through phase angle for participants from CHUM and MUHC (not UAH). Phase angle will be the measure used, representing the ratio of resistance to reactance, as an angle. This is part of the nutrition assessment/overall nutrition status.
Concentration of serum phosphorus (mmol/L) | At baseline, post-induction phase (12 weeks), at 6 months, at 8 months, at 3-month post-transplant.
  At the end of the study, biochemistry will be retrospectively obtained from the participant's medical chart for those occurring within 2 weeks of the scheduled assessment dates found below:
Concentration of serum potassium (mmol/L) | At baseline, post-induction phase (12 weeks), at 6 months, at 8 months, at 3-month post-transplant.
  At the end of the study, biochemistry will be retrospectively obtained from the participant's medical chart for those occurring within 2 weeks of the scheduled assessment dates found below:
Percentage of serum A1C | At baseline, post-induction phase (12 weeks), at 6 months, at 8 months, at 3-month post-transplant.
  At the end of the study, biochemistry will be retrospectively obtained from the participant's medical chart for those occurring within 2 weeks of the scheduled assessment dates found below:
Incidence of anxiety as assessed by Generalized Anxiety Disorder Seven-Item Scale (GAD-7) | At baseline, post-induction phase (12 weeks), at 6 months, at 8 months, at 3-month post-transplant.
  Generalized Anxiety Disorder Seven-Item Scale (GAD-7): this is a 7-question self-report questionnaire completed by participants at the timepoints specified below, indicating the possibility of presence of anxiety. The GAD-7 ranges from 0 to 21, with a lower score indicating minimal anxiety, and a higher score indicating severe anxiety.
Incidence of depression as assessed by the Patient Health Questionnaire (PHQ-8) | At baseline, post-induction phase (12 weeks), at 6 months, at 8 months, at 3-month post-transplant.
  Patient Health Questionnaire (PHQ-8); this is an 8-question self-report questionnaire completed by participants at the timepoints specified below, indicating the possibility of presence of depression. The PHQ-8 ranges from 0 to 24, with a higher score indicating worse health outcomes. Specifically, a score of 3-6/6 for the first 2 questions indicates anxiety, and a score of 3-6/6 on the last 2 questions indicates depression. Higher scores indicate indicate increasing severity of anxiety or depression.
Level of safety as assessed by number/severity of recorded adverse events related to the intervention | from recruitment to end of intervention
  All adverse events will be recorded. Upon review by the investigator, adverse events will be categorized by "related to the intervention" or "unrelated to the intervention" and categorized into three categories: musculoskeletal (e.g., pain, fall), cardiovascular or kidney related. Adverse events will be graded in terms of severity (Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening; and Grade 5: Death).
Trends identified in post-transplant recovery trajectory as sourced from electronic medical chart information | at 3-month post-transplant
  Information collected will include (1) intensive care unit length of stay, (2) hospital length of stay, (3) number of readmissions to hospital within 3 months after the surgery, (4) discharge destination, (5) allograft function.
Level of acceptability of the intervention as assessed by quantitative semantic differential scale | Post-induction phase (at 12-weeks), and at 8-months
  Acceptability of the intervention will be assessed in a subset of patients in the intervention group using both quantitative and qualitative data. Quantitative data will include results from a semantic differential scale and from the closed-ended questions of a semi-structured telephone interview (see outcome measure 25). Based on the semantic differential scale, the intervention will be acceptable if a total score of a minimum of 16 is obtained.
Level of acceptability of the intervention as assessed by qualitative author-generated questionnaire | at 8-months
  Acceptability of the intervention will be assessed in a subset of patients in the intervention group using both quantitative and qualitative data. Quantitative data will include results from a semantic differential scale (see outcome measure 23) and from the closed-ended questions of a semi-structured author-generated telephone questionnaire (guided by previous usability/acceptability studies).

CONTACTS AND LOCATIONS:
Overall Officials: Tania Janaudis-Ferreira, PhD, Principal Investigator — Research Institute of McGill University Health Centre (RI-MUHC)
Locations (2):
- Canada (2):
  - Centre de recherche - Centre Hospitalier de l'Université de Montréal (CRCHUM), Montreal, Quebec
  - Research Institute - McGill University Health Centre (RI-MUHC), Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Summary results will be available on the trial registry site within 12 months from the last visit of the last participant.
  Other data will be shared on request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 12 months from the last visit of the last participant.
Access Criteria: Access to anonymized IPD can be requested by researchers.